CLINICAL TRIAL: NCT06368609
Title: Preliminary Evaluation of Two Rapid Diagnostic Test Prototypes for Strongyloides Stercoralis Infection
Acronym: PROTOSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-09
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Strongyloides Stercoralis Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RDT (Rapid Diagnostic Test) arm (Other): The sera will be selected from the database of the Tropica biobank, based on the given exclusion/inclusion criteria.
  The samples will be tested after thawing shortly before the procedures. Each serum sample will be used for running the two RDTs (IgG and IgG4). Two independent readers will report the test results blinded from each other. In case of discrepancies, a third reader will be involved.
  Interventions: Diagnostic Test: IgG RDT; Diagnostic Test: IgG4 RDT

INTERVENTIONS:
Diagnostic Test: IgG RDT — Sera will be thawed at room temperature; 15 µL of serum will be added to the sample pad of each dipstick, which will then be placed upright into a well containing 3 drops of buffer. The pads at the bottom of the dipstick shall then wick up the buffer to run up the nitrocellulose membrane towards the absorbent pad. The results can be read after 15-20 minutes. The presence of the control line will indicate proper execution of the test, with valid result. In case of absence of this line, the result will be considered invalid. Positive results will be defined as test with presence of both control and positive (including faint) lines; negative results will be defined as tests with presence of control line only.
Diagnostic Test: IgG4 RDT — Sera will be thawed at room temperature; 15 µL of serum will be added to the sample pad of each dipstick, which will then be placed upright into a well containing 3 drops of buffer. The pads at the bottom of the dipstick shall then wick up the buffer to run up the nitrocellulose membrane towards the absorbent pad. The results can be read after 15-20 minutes. The presence of the control line will indicate proper execution of the test, with valid result. In case of absence of this line, the result will be considered invalid. Positive results will be defined as test with presence of both control and positive (including faint) lines; negative results will be defined as tests with presence of control line only.

SUMMARY:
Single center, no profit experimental study on sera available in the Tropica Biobank.

ELIGIBILITY:
Inclusion Criteria:

* Serum from immigrants from S. stercoralis endemic countries (i.e. individuals from Africa, Latin America, South-East Asia and western Pacific regions);
* Serum with a matched result of APC and/or PCR for S. stercoralis (i.e. the latter test/s done in the same day or ±30 days from the collection of the serum) and of serology assays (IFAT and/or ELISA) in use in our laboratory.

Exclusion Criteria:

* Unavailable/insufficient quantity of serum
* Serum from individuals who received treatment with ivermectin in the previous 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
RDTs IgG results: positive or negative | baseline
  RDTs (IgG) results will be classified as positive or negative according to the manufacturer instructions. For the composite reference standard definition: a true positive will be defined as at least one positive faecal test result. True negative will be defined as all test results (faecal and serological) being negative.
RDTs IgG4 results: positive or negative | baseline
  RDTs (IgG4) results will be classified as positive or negative according to the manufacturer instructions. For the composite reference standard definition: a true positive will be defined as at least one positive faecal test result. True negative will be defined as all test results (faecal and serological) being negative.

SECONDARY OUTCOMES:
Agreement between readers | baseline
  Agreement between two independent readers of the RDTs results

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy